CLINICAL TRIAL: NCT01155388
Title: A Randomized, Open-Label, Active-Controlled Study of the Safety, Efficacy, and Pharmacokinetics of Ferumoxytol Compared With Oral Iron for the Treatment of Iron Deficiency Anemia in Pediatric Subjects With Nondialysis-dependent Chronic Kidney Disease
Brief Title: A Trial of Ferumoxytol for the Treatment of Iron Deficiency Anemia in Pediatric Participants With Nondialysis-Dependent Chronic Kidney Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Several factors contributed to significant challenges in enrollment and led the Sponsor to discontinue the AMAG-FER-CKD-252 study as designed.
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-CKD-252
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia; Nondialysis-dependent Chronic Kidney Disease
Keywords: Iron deficiency anemia; Feraheme; ferumoxytol; CKD; pediatric; nondialysis-dependent
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; Iron; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferumoxytol (Experimental): Participants will receive 1 of the following 2 ferumoxytol dose regimens:
  * Four IV injections of ferumoxytol 3.5 mg Fe/kg (maximum of 255 mg/dose) administered on nonconsecutive days within a 14-day period as follows: Day 1 (dose 1), Days 3* through 10 (dose 2), Days 5 through 12 (dose 3), and Days 7 through 14 (dose 4). *Participants participating in PK sampling received the second dose on Day 4 after the 72-hour PK sample was collected.
  * Two IV injections of ferumoxytol 7.0 mg Fe/kg (maximum of 510 mg/dose), the first administered on Day 1 and the second on Days 3 through 9.
  Interventions: Drug: Ferumoxytol
- Oral Iron (Active Comparator): Participants will receive oral iron: 2.5 mg Fe/kg twice daily (maximum of 100 mg/dose) on Days 1 through 35.
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Ferumoxytol — Experimental: Ferumoxytol
  Arms: Ferumoxytol
Drug: Oral Iron — Active Comparator: Oral iron
  Other Names: Ferrous fumarate
  Arms: Oral Iron

SUMMARY:
Study evaluating the efficacy and safety of intravenous (IV) ferumoxytol compared with oral iron for the treatment of pediatric participants with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Study AMAG-FER-CKD-252 was a study evaluating the efficacy and safety of IV ferumoxytol in pediatric participants with nondialysis-dependent CKD. Study AMAG-FER-CKD-251 (NCT01155375) was a study evaluating the efficacy and safety of IV ferumoxytol in pediatric participants with dialysis-dependent CKD. Due to significant challenges with enrollment for both studies, Study AMAG-FER-CKD-252 was combined with Study AMAG-FER-CKD-251 and enrollment continued under Study AMAG-FER-CKD-251. The enrollment number (n=14) includes the number of participants for both AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies, combined.

Participants were enrolled by age cohorts in a stepwise manner following a safety review by the Data Safety Monitoring Board of 1 age cohort prior to enrollment of a subsequent age cohort, with progression from oldest to youngest. Randomization was stratified by the following age cohorts: 12 to <18 years, 6 to <12 years, 2 to <6 years, and 6 months to <2 years.

ELIGIBILITY:
Key Inclusion Criteria for this study include:

1. Males or females 6 months to <18 years of age
2. Nondialysis dependent CKD, including kidney transplant recipients
3. Has iron deficiency anemia defined as: a) hemoglobin level <11.0 grams (g)/deciliter (dL) and b) transferrin saturation level <20%
4. Female participants of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to Screening and agree to remain on birth control until completion of participation in the study

Key Exclusion Criteria for this study include:

1. History of allergy to either oral or IV iron
2. Allergy to two or more classes of drugs
3. Female participants who are pregnant, intend to become pregnant, are breastfeeding, within 3 months postpartum, or have a positive serum/urine pregnancy test
4. Hemoglobin level ≤7.0 g/dL
5. Serum ferritin level >600 nanograms/milliliter

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-10-17 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AMAG Pharmaceuticals, Inc., Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to significant challenges with enrollment for both studies, Study AMAG-FER-CKD-252 was combined with Study AMAG-FER-CKD-251 (NCT01155375) and enrollment continued under Study AMAG-FER-CKD-251. Data is for the combined Study AMAG-FER-CKD-252 and Study AMAG-FER-CKD-251.The results for the combined studies are included in this record.
Groups:
- Ferumoxytol: Participants received 1 of the following 2 ferumoxytol dose regimens:
  * Four intravenous (IV) injections of ferumoxytol 3.5 milligrams (mg) iron (Fe)/kilogram (kg) (maximum of 255 mg/dose) administered on nonconsecutive days within a 14-day period as follows: Day 1 (dose 1), Days 3* through 10 (dose 2), Days 5 through 12 (dose 3), and Days 7 through 14 (dose 4). *Participants participating in pharmacokinetic (PK) sampling received the second dose on Day 4 after the 72-hour PK sample was collected.
  * Two IV injections of ferumoxytol 7.0 mg Fe/kg (maximum of 510 mg/dose), the first administered on Day 1 and the second on Days 3 through 9.
- Oral Iron: Participants received oral iron 2.5 mg Fe/kg twice daily (maximum of 100 mg/dose) on Days 1 through 35.
Period: Overall Study
Arm/Group | Ferumoxytol | Oral Iron
Started (Data are for the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies.) | 8 | 6
Received at Least 1 Dose of Study Drug | 8 | 6
Completed | 7 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population is defined as participants who received any amount of study drug. Data are for the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies. The safety analysis is based on actual treatment received.
Groups:
- Ferumoxytol: Participants received 1 of the following 2 ferumoxytol dose regimens:
  * Four IV injections of ferumoxytol 3.5 mg Fe/kg (maximum of 255 mg/dose) administered on nonconsecutive days within a 14-day period as follows: Day 1 (dose 1), Days 3* through 10 (dose 2), Days 5 through 12 (dose 3), and Days 7 through 14 (dose 4). *Participants participating in PK sampling received the second dose on Day 4 after the 72-hour PK sample was collected.
  * Two IV injections of ferumoxytol 7.0 mg Fe/kg (maximum of 510 mg/dose), the first administered on Day 1 and the second on Days 3 through 9.
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Oral Iron | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.65) | 13.8 (4.52) | 14.6 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change In Hemoglobin From Baseline To Week 5
Description: Mean changes in hemoglobin from Baseline to Week 5 were to be presented. Despite efforts to complete the studies as designed, several factors contributed to significant challenges in enrollment and led the sponsor to discontinue the combined AMAG FER-CKD-252 and AMAG FER-CKD-251 studies. Blood samples were collected, but not run through an analysis to obtain outcome measure data. As such, the data set for this primary outcome measure cannot be summarized nor can the statistical analysis, as described in the protocol, be provided in a way that will provide any significant data based upon the limited study datasets.
Time Frame: Baseline, Week 5
Population: Intent-to-Treat Population included all randomized participants who had received at least 1 dose of study drug. Sample data were collected, but not run through any analysis to obtain outcome measure data. As such, summary of the data set is not possible.
Arm/Group | Ferumoxytol | Oral Iron
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Area Under The Curve Of Ferumoxytol
Description: Ferumoxytol concentrations were to be determined using a drug-specific nuclear magnetic resonance assay. Blood samples were to be collected at specified times predose and postdose at the time of the first dose from 6 participants in each age-dose group. Sampling for participants <6 years of age will be minimized to the fewest number of time points required for population PK analysis based on preliminary PK data from the first 2 age cohorts. Blood samples were collected, but not run through an analysis to obtain outcome measure data. As such, the data set for this secondary outcome measure cannot be summarized in a way that will provide any significant data based upon the limited study datasets.
Time Frame: Baseline; 10, 30, 120, and 360 minutes postdose; 24, 48, and 72 hours postdose
Population: The PK population included all randomized participants who received at least 1 dose of study drug and consented to PK sampling. Sample data were collected, but not run through any analysis to obtain outcome measure data. As such, summary of the data set is not possible.
Arm/Group | Ferumoxytol | Oral Iron
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Randomization up to 7 weeks (Follow-up)
Description: Due to significant challenges with enrollment for both studies, Study AMAG-FER-CKD-252 was combined with Study AMAG-FER-CKD-251 and enrollment continued under Study AMAG-FER-CKD-251. The adverse events for the combined studies are included in this record.
Arm/Group | Ferumoxytol | Oral Iron
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6
Other Adverse Events (participants affected / at risk) | 6/8 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=8) | Oral Iron (N=6)
Acute gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=8) | Oral Iron (N=6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ventricular flutter (Cardiac disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Residual urine volume decreased (Investigations) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
While sample data were collected, it was not run through any analysis to obtain the necessary outcome measure data. As such, summary of the data set is not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data has been received by Sponsor, the Site and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 120 days to allow Sponsor to protect its interests.